CLINICAL TRIAL: NCT07281599
Title: Evaluation of the Q-Pad hrHPV Test System for Identifying Precancer
Acronym: EQUIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qurasense (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ALM_QT2/DOC-392
Record Dates: First submitted 2025-12-03; First posted 2025-12-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: HPV Infection; HPV 16 Infection; High Risk HPV; Cervical Cancer Screening; Cervical Cancer Cin Grade; Cervical Cancer (Early Detection); HPV; HPV (Human Papillomavirus)-Associated; HPV DNA; HPV Infections; Screening Test
Keywords: Q-Pad; Self-sampling; Self-collection; self-collect; cervical cancer screening; menstural blood; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Genital Diseases; Papillomavirus Infections; HPV; high risk HPV; pap smear; at-home collection
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Genital Diseases | interventions — Colposcopy

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, single-cohort, paired-sample diagnostic accuracy study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Non-invasive, passive self-collection / Clinician collection (Other): Participants referred for colposcopy after abnormal cervical screening will collect menstrual blood at home using the Q-Pad kit and mail the sample for hrHPV testing. At the colposcopy visit, they will have a clinician-collected cervical specimen obtained for hrHPV testing and undergo colposcopy with biopsy as part of standard care.
  Interventions: Device: Q-Pad hrHPV Test System

INTERVENTIONS:
Device: Q-Pad hrHPV Test System — Participants will receive a mailed Q-Pad Kit, which includes two Q-Pads (menstrual pads with removable collection strips called Q-Strips), a Q-Strip Container with desiccant for storing and shipping the strips, and a prepaid return mailer. During the menstrual cycle after their colposcopy visit, participants will follow the Instructions for Use to passively collect menstrual blood with the Q-Pads, then remove the Q-Strips and place them in the Q-Strip Container for mailing to the central laboratory for hrHPV testing. At the colposcopy visit, the clinician will also collect a cervical sample in ThinPrep liquid-based cytology medium for hrHPV testing, which will serve as the comparator specimen.
  Other Names: Q-Pad Kit; Colposcopy; Clinician collection

SUMMARY:
The EQUIP Study is testing whether high-risk human papillomavirus (hrHPV), the virus that causes most cervical cancers, can be accurately detected from menstrual blood collected at home. People who have been referred for colposcopy after an abnormal Pap or hrHPV test will use the Q-Pad Kit during their period to collect menstrual samples on a special menstrual pad and mail them to a central laboratory for hrHPV testing.

The same participants will have a standard cervical sample collected for routine hrHPV testing and will undergo colposcopy as part of their usual care. By comparing hrHPV results from menstrual samples with results from cervical samples and biopsy findings, the study will evaluate how well the Q-Pad hrHPV Test System detects cervical precancer and will also assess how easy and acceptable it is for participants to use this at-home collection method.

DETAILED DESCRIPTION:
The EQUIP Study is a prospective, multicenter method-comparison study designed to evaluate the diagnostic performance of the Q-Pad hrHPV Test System for cervical cancer screening. Menstruating adults referred for colposcopy after an abnormal cervical screening result receive a mailed Q-Pad Kit and use it during the menstrual cycle immediately after their clinic visit to collect a menstrual samples at home, guided by written instructions and an optional accompanying smartphone application. These samples are returned by mail to a central laboratory, where hrHPV testing is performed using a PCR assay.

At the colposcopy visit, clinicians obtain a standard cervical specimen for routine cytology and hrHPV testing on the same assay platform and perform colposcopy with biopsy as clinically indicated. Each participant therefore provides both an at-home menstrual sample (index test) and a clinician-collected cervical sample (comparator) within the same episode of care, with biopsy and histopathology providing disease status. The study focuses on comparing hrHPV results between the two specimen types and on evaluating safety, specimen adequacy, and participant usability and acceptability of the Q-Pad at-home menstrual collection approach.

ELIGIBILITY:
Inclusion Criteria:

* You are 25 years old or older and have an intact cervix.
* You were referred for a colposcopy after an abnormal Pap or HPV screen.
* Your periods come regularly-about every 21-35 days.
* You own a smartphone, have an email address, and can read the Qvin app instructions in English.
* You are willing to sign the consent form (electronically).
* You agree to use a condom for any vaginal intercourse or shared penetrative toy use from Q-Pad collection until the colposcopy visit if engaging with a new sexual partner during this period.

Exclusion Criteria:

* You are pregnant or think you might be.
* You are unwilling or unable to use the two Q-Pads and mail them back (mailing costs are covered).
* You had treatment for cervical pre-cancer (CIN2+)-such as LEEP, cone, or ablation-within the last 12 months.
* You have already joined this study or are in another cervical-screening / HPV study right now.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Clinical Performance vs Histology | Through study completion, an average of 1 year.
  Clinical sensitivity defined as the proportion of participants with biopsy-confirmed CIN2+ whose menstrual-blood hrHPV result (Q-Pad hrHPV Test System) is positive and Clinical specificity defined as the proportion of participants with <CIN2 on histology whose menstrual-blood hrHPV result is negative.
Proportion of participants with at least one reportable device-related adverse event (ADE or SADE) | Through study completion, an average of 1 year.
  Proportion of participants who experience at least one adverse event or device deficiency that is not on the protocol's non-reportable event list.

SECONDARY OUTCOMES:
Positive, negative, and overall percent agreement between Q-Pad hrHPV testing and clinician-collected cervical hrHPV testing | Through study completion, an average of 1 year.
  Positive percent agreement (PPA), negative percent agreement (NPA), and overall percent agreement (concordance) between the Q-Pad hrHPV Test System result on menstrual blood (index test) and the hrHPV result from the paired clinician-collected cervical ThinPrep specimen (comparator test).
Q-Pad hrHPV Test System validity rate and participant usability/acceptability | Through study completion, an average of 1 year.
  Proportion of returned Q-Pad menstrual collections that yield a valid hrHPV test result in the central laboratory (i.e., not invalid or quantity-not-sufficient [QNS]), together with participant usability and acceptability scores for the Q-Pad kit.

OTHER OUTCOMES:
CIN3+ Clinical Sensitivity & Specificity | Through study completion, an average of 1 year.
  Using biopsy as reference, calculate clinical sensitivity/specificity of Q-Pad hrHPV for detecting CIN3+ lesions

CONTACTS AND LOCATIONS:
Overall Officials: Paul Blumenthal, MD, MPH, Study Director
Locations (4):
- United States (4):
  - Planned Parenthood of Southern New England, New Haven, Connecticut
  - Planned Parenthood North Central States, Minneapolis, Minnesota
  - Planned Parenthood of Greater Ohio (PPGOH), Akron, Ohio
  - Planned Parenthood Association of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arbyn M, Peeters E, Benoy I, Vanden Broeck D, Bogers J, De Sutter P, Donders G, Tjalma W, Weyers S, Cuschieri K, Poljak M, Bonde J, Cocuzza C, Zhao FH, Van Keer S, Vorsters A. VALHUDES: A protocol for validation of human papillomavirus assays and collection devices for HPV testing on self-samples and urine samples. J Clin Virol. 2018 Oct;107:52-56. doi: 10.1016/j.jcv.2018.08.006. Epub 2018 Aug 22. PMID 30195193
- [Background] Naseri S, Young S, Cruz G, Blumenthal PD. Screening for High-Risk Human Papillomavirus Using Passive, Self-Collected Menstrual Blood. Obstet Gynecol. 2022 Sep 1;140(3):470-476. doi: 10.1097/AOG.0000000000004904. Epub 2022 Aug 3. PMID 35926207
- [Background] U.S. Food and Drug Administration, "510(k) Substantial Equivalence Determination Decision Summary: Q-Pad A1c Test System (K231465)," 2023, accessed June 11, 2025, https://www.accessdata.fda.gov/cdrh_docs/pdf23/K231465.pdf.
- See also: Qurasense, Inc. DBA Qvin public facing website — https://www.qvin.com